CLINICAL TRIAL: NCT05838300
Title: Lexion AP 50/30 Warmed Humidified Real Time CO2 Insufflation vs Airseal Recirculated CO2/Air Insufflation in Minimally Invasive Bariatric (Gastric Bypass) Surgery: A Randomized Controlled Study of Clinical Evaluation
Brief Title: Lexion AP 50/30 Warmed Humidified Real Time CO2 Insufflation vs Airseal Recirculated CO2/Air Insufflation in Minimally Invasive Bariatric (Gastric Bypass) Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Erik B Wilson, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC-MS-22-0444
Record Dates: First submitted 2023-04-04; First posted 2023-05-01 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Bariatric Surgery
Keywords: carbon dioxide; minimally invasive surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Warm humidified CO2 (Experimental)
  Interventions: Device: Warm humidified CO2
- Dry CO2 (Active Comparator)
  Interventions: Device: Dry CO2

INTERVENTIONS:
Device: Warm humidified CO2 — Participants will receive warm (37°C) and humidified (95%) CO2.The humidification and warming device to be used is AlwaysPneumo® AP 50/30 InsuflowPort® (Lexion Medical, FDA approved) which is a specialized port that delivers warmed (95° F) and humidified (95% relative humidity) CO2, the source of which is a standard CO2 tank or wall source
  Arms: Warm humidified CO2
Device: Dry CO2 — Participants will receive standard cold (19-21 °C) and non-humidified (0%) CO2 insufflation with Airseal Insufflator
  Arms: Dry CO2

SUMMARY:
The purpose of this study is to To determine the effect of warm and humidified (WH) carbon dioxide (CO2) on post-operative pain/analgesia requirement in patients undergoing laparoscopic bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective bariatric primary or revision procedures and hiatal hernia repair procedures for all indications.

Exclusion Criteria:

* emergency surgery, reoperation within 30 days
* patients who are taking pain medications (narcotics) daily preoperatively for whatever reason
* history of narcotics addiction
* paraplegic and quadriplegic patients
* dementia or altered mental status
* patients on steroids
* pregnant women
* psychiatric patients
* minors
* unable to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain as assessed by the visual analog scale (VAS) | First 24 hours after surgery
  This will be measured as a binary outcome variable (pain will be determined as VAS >/= 4, and no pain will be VAS < 4). This will be determined on post-operative day 1 as an average of the two pain scores.

SECONDARY OUTCOMES:
Intraoperative temperature measured via bladder probe (average of the measurements on the anesthesia record) | From the start surgery to the end of the surgery in minutes
  the body temperature of the patient from the bladder
Temperature in the PACU | From the time the patient enters PACU to the time patient leaves the PACU in minutes
  the temperature of the patient in PACU measured each 30 minutes in PACU
Analgesic requirements in the Post Anesthesia Care Unit (PACU) | From the time the patient enters the PACU to the time patient leaves the PACU in minutes
  the amount, type and doses of drugs administered in the PACU to the patient
Volume of CO2 consumed during the procedure | from the time the CO2 machine is turned on to the time the CO2 machine is turned off in minutes
  the amount/volume of CO2 used during the procedure
Length of hospital stay | the amount of hours the patient stays in the hospital (ie 24 hours)
  from admission to the hospital to discharge from the hospital in hours
Duration of surgery | From start of the surgery to the end of the surgery in minutes
  from the start of the first incision of surgery to the closing of the last incision of surgery in minutes
Incision length | measurement in centimeters the patients incision lengths at the closing of the surgery
  the length of the incisions on the patient abdomen
Intra-operative and total hospital costs | from the admission to discharge of the patient in hours
  the cost for the intra-operative services and total hospital hospital costs
Total narcotic use intra-operatively (in morphine milliequivalents) | volume of narcotics used from the beginning of surgery to end of surgery in milliequivalents
  volume of narcotics used during the operation
Postoperative Analgesia Requirement measured in morphine milliequivalents | any postoperative analgesia used after the surgery is completed to the discharge of the patient from the hospital
  the amount of analgesia used type, dose and amounts used post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Erik Wilson, MD, FACS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No